CLINICAL TRIAL: NCT00143195
Title: Open Label Study Comparing Amlodipine vs Long-acting Nitrates in Patients With Chronic Stable Angina.
Brief Title: Amlodipine vs Nitrates Study in Patients With Chronic Stable Angina
Acronym: ANISSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0531076
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia | interventions — Amlodipine; Isosorbide; Hematologic Tests; Exercise Test

INTERVENTIONS:
Drug: Amlodipine
Drug: iso- 5 - mononitrate
Procedure: Blood tests
Procedure: Exercise Stress Test

SUMMARY:
The objective of study is to compare the anti-ischemic efficacy and safety profiles of once daily amlodipine or isosorbide-5-mononitrate in the treatment of stable asymptomatic and symptomatic myocardial ischemia

ELIGIBILITY:
Inclusion Criteria:

* Outpatients > =18 years of age with diagnosed clinically stable angina pectoris

Exclusion Criteria:

* Patients with congestive heart failure, clinically significant cardiovascular disease, standing systolic blood pressure of less than 100mmHg, concomitant anti-anginal therapies similar to sublingual NTG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2001-04; Study Completion 2005-01

PRIMARY OUTCOMES:
Evaluate the time to 1mm ST depression

SECONDARY OUTCOMES:
The number of patients experiencing angina attacks The frequency of hospitalizations due to angina attacks Time to onset of 1mm ST segment depression Total external workload performed Safety

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Greece (10):
  - Pfizer Investigational Site, Athens, Attica
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Holargos/Athens
  - Pfizer Investigational Site, Loannina
  - Pfizer Investigational Site, N. Ionia
  - Pfizer Investigational Site, Pátrai
  - Pfizer Investigational Site, Rio, Patra
  - Pfizer Investigational Site, Thessaloniki
  - Pfizer Investigational Site, Voula/Athens
  - Pfizer Investigational Site, Zakynthos

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0531076&StudyName=Amlodipine+vs+NItrates+Study+in+Patients+with+Chronic+Stable++Angina+%28ANISSA%29